CLINICAL TRIAL: NCT02846701
Title: DULOPLASM Study: Pilot Study on Mechanisms of Analgesic Action of Duloxetine: Effective Dosage of Duloxetine at the Peak and at the Lowest Plasma Concentrations
Brief Title: Determination of the Antidepressant Duloxetine in Plasma to Improve the Knowledge of the Analgesic Action of Antidepressants on Chronic Neuropathic Pain
Acronym: DULOPLASM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6314
Record Dates: First submitted 2016-07-01; First posted 2016-07-27 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; Antidepressant; Duloxetine; Liquid Chromatography; Mass Spectrometry
MeSH Terms: conditions — Neuralgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient treated by duloxetine (Other)
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — The concentration of duloxetine is measured by liquid chromatography coupled to tandem mass spectrometry on blood sample

SUMMARY:
The primary purpose of this protocol is to evaluate the lowest plasma concentration (ie before the daily taking dose of duloxetine) in patients relieved of at least 30% of their neuropathic pain with duloxetine treatment.

The secondary purpose of this protocol is to determine plasmatic concentration peak (ie 6 hours after taking duloxetine) in patients relieved of at least 30% of their neuropathic pain with duloxetine treatment.

Others secondary purposes are to evaluate the intensity of neuropathic pain, to assess the degree of pain relief and to evaluate the sensation of the global improvement experienced by the patient.

ELIGIBILITY:
Inclusion criteria:

* aged 40 to 75 years old
* relieved of their neuropathic pain by 60 mg of duloxetine treatment (with a differential of> 30% in the intensity of neuropathic pain with NRS, before and after treatment initiation)

Exclusion criteria:

* concomitant treatment with enoxacin, fluvoxamine, flecainide, propafenone, metoprolol, risperidone, verapamil, omeprazole, modafinil, mequitazine, propafenone, tamoxifen, Monoamine Oxidase Inhibitors.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Measurement of the lowest plasma concentration of duloxetine in pmol/mL. | The concentration of duloxetine is measured by liquid chromatography coupled to tandem mass spectrometry on blood sample taken at the inclusion visit (V0), before the daily morning dose of duloxetine.

SECONDARY OUTCOMES:
Measurement of the plasma concentration peak of duloxetine in pmol/mL. | The concentration of duloxetine is measured by liquid chromatography coupled to tandem mass spectrometry on blood sample taken during the V1 visit (28 days after V0, 6 hours after the daily morning dose of duloxetine).

OTHER OUTCOMES:
Intensity of his pain assessed by Numeric Rating Scale (NRS) in 11 points. | at inclusion visit V0 and at V1 visit (28 days after the inclusion visit V0).
  The patient will daily report the intensity of his pain on a Numeric Rating Scale (NRS) in 11 points. The mean intensity of pain is measured at V0 and V1 visits.
Sensation of improvement | at inclusion (V0 visit)
  The sensation of improvement experienced by the patient is assessed at V0 visit on a patient's global impression of change (PGIC) in 7 points scale.

IPD SHARING:
Plan to Share IPD: No